CLINICAL TRIAL: NCT06237777
Title: An Open, Dose-escalation Clinical Study Evaluating the Safety, Tolerability and Initial Efficacy of SKG0106 Intravitreal Injection in Diabetic Macular Edema (DME) Patients in China
Brief Title: A Clinical Study Evaluating the Safety, Tolerability and Initial Efficacy of SKG0106 Intravitreal Injection in Diabetic Macular Edema (DME) Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wang Min (Other)
Collaborators: Lanyue Biotech (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Wang Min, Chief physician, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKG0106-002
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Macular Edema
Keywords: DME

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation (Experimental): SKG0106 one-time deliver
  Interventions: Genetic: SKG0106 intravitreal injection dose level 1, 2 or 3

INTERVENTIONS:
Genetic: SKG0106 intravitreal injection dose level 1, 2 or 3 — SKG0106 is a recombinant adeno-associated virus (rAAV) vector-based in vivo gene therapeutic product.
  Other Names: SKG0106

SUMMARY:
This is a clinical study to evaluate the safety, tolerability and initial efficacy of SKG0106 intravitreal injection in diabetic macular edema (DME) patients.

DETAILED DESCRIPTION:
This is an open, dose-escalation clinical study to evaluate the safety, tolerability and initial efficacy of SKG0106 intravitreal injection in diabetic macular edema (DME) patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to all assessments.
* Age ≥18 years at screening.
* Type 1 or type 2 diabetes mellitus at screening.
* Study eye criteria:

  * Decreased visual acuity attributable primarily to DME.
  * DME involves the macular center.

Exclusion Criteria:

* Active proliferative diabetic retinopathy in the study eye.
* Any current or previous ocular disease in the study eye other than DME that could interfere with macular evaluation or affect central vision at screening or baseline.
* Any active intraocular or periocular infection or active intraocular inflammation of the study eye at screening or baseline.
* History of idiopathic or autoimmune uveitis in the study eye at screening or baseline.
* Prior gene therapy in either eye.
* History of vitreoretinal surgery in the study eye.
* Uncontrolled blood pressure at screening or baseline defined as systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg.
* History of treated or untreated malignancy of any organ system within the past 5 years.
* Pregnant or lactating women.
* Women of reproductive age, defined as all women who are biologically capable of being pregnant, unless they use highly effective contraceptive methods between the time of study drug administration and 3 months after EOS (end of study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Type, severity, and incidence of ocular and systemic AEs | AEs: Adverse Events
  48 weeks
Incidence of DLT | 4 weeks
  DLT (Dose-limiting Toxicity) is judged by assessing the following AEs such as:
  * Severe visual acuity decline
  * Endoophthalmitis by investigator
  * Vitreous hemorrhage by investigator

SECONDARY OUTCOMES:
Mean change from baseline in BCVA | 48 weeks
  BCVA (Best Corrected Visual Acuity) of the study eye is examined by the Early Treatment of Diabetic Retinopathy Study (ETDRS) testing.
Mean change from baseline in CST | 48 weeks
  CST (Central Subfield Thickness) is measured by Spectral domain optical coherence tomography (SD-OCT).
Mean change from baseline in patient-reported outcome (VFQ-25) scale score | 48 weeks
  Both the total scale and subscale scores of the VFQ-25 (25-Item Visual Function Questionnaire) is ranging from 0 to 100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Min Wang, Doctor, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Eye & ENT Hospital of Fudan University, Shanghai